CLINICAL TRIAL: NCT04810221
Title: Postmarket Clinical Follow-up Study (PMCF) to Confirm the Performance of the Wearable Pulse-Oximeter BrOxy M
Brief Title: Postmarket Clinical Follow-up Study to Confirm the Performance of the Wearable Pulse-Oximeter BrOxy M (SOMBRERO)
Acronym: SOMBRERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life Meter srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01M2020-CH.LMD
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-02

CONDITIONS: Laboratory Testing on Healthy Volunteers to Verify SpO2 and Heart Rate (HR) Accuracy of BrOxy M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Measure of SpO2 and HR obtained in enrolled subjects using BrOxy M and a reference pulse oximeter in paired observations
  Interventions: Other: Controlled desaturation study

INTERVENTIONS:
Other: Controlled desaturation study — Measure of SpO2 and Heart Rate by BrOxy M device and reference device in a controlled desaturation study.

SUMMARY:
This study is a post market clinical follow up study performed to confirm the performance of BrOxy M pulse oximeter in comparison with a reference, CE marked, pulse oximeter equipment in a controlled desaturation study over a range between 80% and 100% peripheral oxygen saturation (SpO2).

The study will be performed on a group of healthy volunteers in a controlled clinical setting.

DETAILED DESCRIPTION:
This study is a post market clinical follow up study performed to confirm the performance of BrOxy M pulse oximeter in comparison with a reference, CE marked, pulse oximeter equipment (Nellcor™ Bedside Respiratory Patient Monitoring System model PM1000N, Covidien LLC, USA) in a controlled desaturation study over a range between 80% and 100% SpO2.

The study will be performed on a group of healthy volunteers in a controlled clinical setting. Due to the use of a controlled desaturation protocol foreseen by the standard ISO 80601-2-61:2017, this study is classified as an interventional post-market clinical study in accordance with Annex I of EN ISO 14155:2020.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects of both sexes with an age ≥ 18 and ≤ 50.
2. American Society of Anesthesiology (ASA) classification 1
3. Positive Allen's test
4. Intact and healthy skin on the selected wrist
5. Wrist circumference diameter between 150 mm e 200 mm.
6. Normal electrocardiogram (ECG) obtained at screening or within 2 months prior to screening
7. Ability to understand and execute the required study procedures and provide an informed consent to the study

Exclusion Criteria:

1. Presence of at least one of the following altered hemoglobin parameters at screening:

   1. Alpha-hemoglobin (αHb) ≤ 10 gr/dl
   2. Carboxy-hemoglobin (COHb) ≥ 3%
   3. Methaemoglobin (MetHb) ≥ 2%
2. For pre-menopausal female subjects only: positive pregnancy test performed at screening on urines or capillary blood
3. Presence of any cardiovascular pathology in medical history.
4. Any episodes of respiratory infection during the 30 days prior to screening
5. Any prior experience of Dyspnea
6. Hospitalization during the 2 months prior to screening, for any reason.
7. Chronic drug intake known to interfere with gaseous exchanges or induce changes in cardiac frequency
8. Presence of any medical condition not allowing the subject to perform the required test
9. Known allergy to adhesive tapes
10. Participation in an interventional study with a medicinal product or a medical device in the 30 days prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Marinari, Medicine, Principal Investigator — Ospedale "SS. Annunziata", Via dei Vestini, 66100 Chieti, Italy
Locations (1):
- Ospedale "SS. Annunziata", Chieti, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 19 subjects signed the informed consent and were screened for participating in the study. Of these, 3 subjects were smokers with carboxyhemoglobin (COHb) ≥ 3% and were considered screen failures. The remaining 16 were eligible and were enrolled.
Groups:
- Experimental: Measure of peripheral oxygen saturation (SpO2) and heart rate (HR) obtained in enrolled subjects using BrOxy M and a reference pulse oximeter in paired observations
Period: Overall Study
Arm/Group | Experimental
Started | 16
Completed | 13 (Included in the 13 subjects which completed the study, it is necessary to consider the case "0", a pilot test for the verification of study procedures. Data from this subject were not used in the statistical evaluation, which therefore included data from 12 eligible subjects that completed the study.)
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: SpO2and HR paired measurements were obtained in parallel from the reference device and BrOxy M.
  The final number of data pairs included in the statistical analyses was 219.
Groups:
- Experimental: Measure of SpO2 and heart rate (HR) obtained in enrolled subjects using BrOxy M and a reference pulse oximeter in paired observations
Arm/Group | Experimental
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Skin pigmentation [Count of Participants; unit: Participants] — Black or white skin
  Participants
    Skin black | 4
    skin white | 8
Body/Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of SpO2 Measurement at 80-100% SpO2
Description: Accuracy of SpO2 measurements obtained with BrOxy M in comparison with the reference pulse oximeter in paired observations over a range between 80% and 100% SpO2. Based on the standard ISO 80601-2-61:2017, the accuracy is stated in terms of the root-mean-square difference between the readings of the BrOxy M and the standard readings of the reference pulse oximeter.
Time Frame: The measures started around 2 minutes after beginning of the test session and ended around 33 minutes later.
Measure: Mean (95% Confidence Interval); unit: A(RMS) - %
Groups:
- Experimental: Controlled desaturation study: Measure of SpO2 and Heart Rate by BrOxy M device and a reference device in a controlled desaturation study, in paired observations.
Arm/Group | Experimental
Number analyzed (Participants) | 12
A(RMS) - % | 2.7 [-5.1 to 5.5]
Statistical Analysis 1: Comparison: Experimental; Test type: Other — Paired T-test 0; p = 0.31, Paired T-test 0; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.17 to 0.54]; Additional statistical analysis were: Bland Altman plot and linear regression analysis

2. Primary Outcome: Accuracy of Heart Rate Measurement at 80-100% SpO2
Description: Accuracy of measurements obtained with BrOxy M with that obtained with the reference pulse oximeter in paired observations. Based on the standard ISO 80601-2-61:2017, the accuracy is stated in terms of the root-mean-square difference between the readings of the BrOxy M and the standard readings of the reference pulse oximeter.
Time Frame: The test started around 2 minutes after beginning of the test session and ended after around 33 minutes.
Measure: Mean (95% Confidence Interval); unit: bpm
Arm/Group | Experimental
Number analyzed (Participants) | 12
bpm | 3.7 [-7.1 to 7.7]
Statistical Analysis 1: Comparison: Experimental; Test type: Other — Paired T test 0; p = 0.32, Paired T test 0; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.24 to 0.75]; Additional statistical analysis were: Bland Altman plot and linear regression analysis

3. Secondary Outcome: Agreement Between Broxy M and Reference Device SpO2 Measurements - Cut Off at 94% SpO2
Description: Cohen's kappa coefficient to evaluate the agreement between Broxy M and the reference device for 94% SpO2 cut off. Cohen's kappa coefficient takes into account the possibility of agreement occurring by chance.
Time Frame: Around 5 min after beginning of the test session
Measure: Number; unit: Cohen's kappa coefficient
Arm/Group | Experimental
Number analyzed (Participants) | 12
Cohen's kappa coefficient | 0.79

4. Secondary Outcome: Agreement Between Broxy M and the Reference Device SpO2 Measurements - Cut Off at 90% SpO2
Description: Cohen's kappa coefficient to evaluate the agreement between Broxy M and the reference device for 90% SpO2 cut off
Time Frame: After around 10 min after beginning of the test session
Measure: Number; unit: Cohen's kappa coefficient
Units Other Than Participants: data pairs
Arm/Group | Experimental
Number analyzed (Participants) | 12
Number analyzed (data pairs) | 219
Cohen's kappa coefficient | 0.80

ADVERSE EVENTS:
Time Frame: The reporting period for adverse events was from the day the subject performed screening examinations until study exit (ie around 1-2 days).
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT04810221/Prot_SAP_000.pdf